CLINICAL TRIAL: NCT02157129
Title: LipoAerosol© Inhalation to Maintain the Functional Integrity of the Tracheo-bronchial System in Patients After Tracheostomy
Brief Title: LipoAerosol© Inhalation After Tracheostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HNO-TUM-LT1
Record Dates: First submitted 2014-05-27; First posted 2014-06-05 (Estimated); Last update posted 2022-07-06 (Actual); Status verified 2017-08

CONDITIONS: Other Tracheostomy Complication
Keywords: Tracheostomy; inflammation; mucous congestion; inhalation therapy; phospholipids
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LipoAerosol© (Experimental): LipoAerosol© inhalation, 5x/d for 30min
  Interventions: Device: LipoAerosol© inhalation
- Physiologic saline inhalation (Other): Physiologic saline inhalation, 5x/d for 30min
  Interventions: Other: Physiologic saline inhalation

INTERVENTIONS:
Device: LipoAerosol© inhalation — LipoAerosol© inhalation, 5x/d for 30min
  Arms: LipoAerosol©
Other: Physiologic saline inhalation — Physiologic saline inhalation, 5x/d for 30min
  Arms: Physiologic saline inhalation

SUMMARY:
Patients after tracheostomy represent a substantial part in the ear nose throat clinic. Long-term intubated patients in intensive care units also profit from tracheostomy due to an improved respiratory toilet. However, after tracheostomy patients demonstrate shunt ventilation bypassing the sinonasal and pharyngeal system. The physiological moistening, cleaning and warming of the breathing air fail resulting in a respiratory inflammation. Beside a variety of supportive medical devices no general recommendation exists at present. Recently, we demonstrated the beneficial application of local phospholipids in Sjoegren's syndrome and antineutrophil cytoplasmatic antibody associated sinonasal vasculitis.

In the current monocentric, two-armed, double-blinded, randomized parallel group study we would like to evaluate the beneficial application of LipoAerosol© when compared with standard physiologic saline inhalation. LipoAerosol© is a licensed, tradable medical device and will be applied as part of its intended use. Liposomal inhalation solution provides moistening, cleaning and warming of the upper and lower respiratory tract and supports the natural moistening film in airway irritations and diseases.

Blood parameter (leucocytes and c reactive protein) and tracheobronchial secretion (Lymphocyte subpopulation, c reactive protein, lactate dehydrogenase, granulocyte macrophage colony stimulating factor, interferon γ, interleukins 10, 12 (p70), 13, 1β, 2, 4, 5, 6, 7, 8, tumor necrosis factor α) will be collected 1, 3, and 10 days after tracheostomy. In addition, medical examination records the number of suction maneuver (0 points: none; 1 point: 5-10x/d; 2 points: 10-20x/d; 3 points: >20x/d), flexible-optical assessment of tracheo-bronchial redness (0 point: none; 1 point: peristomal; 2 points: tracheal; 3 points: tracheo-bronchial) and flexible-optical assessment of mucous congestion (0 point: none; 1 point: fluent; 2 points: tenacious; 3 points: barky).

Subjective estimation of the respiratory impairment will be analyzed via visual analogue scale (Subjective overall impairment, coughing frequency, breathlessness, mucous congestion, color of sputum, consistency of sputum). The study is designed without any additional invasive or incriminating clinical examination.

Aim of the study is to maintain the functional integrity of the tracheo-bronchial system after tracheostomy using LipoAerosol© resulting in a general therapeutic recommendation.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≤24h after tracheostomy and regular patient's consent

Exclusion Criteria:

* No regular patient's consent
* Known allergy for ingredients
* Patients >24h after tracheostomy
* Patients with acute or imminent sepsis
* Patients with existing bronchopulmonary inflammation
* Patients with immunosuppressive therapy
* Patients with poorly adjusted pulmonary disease
* Patients with chronic respiratory insufficiency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Changes in tracheal interleukin 6 levels | at day 10 after tracheostomy
  Tracheal secretion: Interleukin 6

SECONDARY OUTCOMES:
Changes in the number of suction maneuver, tracheo-bronchial redness, and mucous congestion | at day 10 after tracheostomy
  Changes in the respiratory impairment due to the medical estimation at day 10. The medical estimation includes number of suction maneuver (0 points: none; 1 point: 5-10x/d; 2 points: 10-20x/d; 3 points: >20x/d), flexible-optical assessment of tracheo-bronchial redness (0 point: none; 1 point: peristomal; 2 points: tracheal; 3 points: tracheo-bronchial) and flexible-optical assessment of mucous congestion (0 point: none; 1 point: fluent; 2 points: tenacious; 3 points: barky).

OTHER OUTCOMES:
Changes in the inflammatory blood and tracheal secretion parameters | at day 1, 3, 10 after tracheostomy
  Blood: C reactive protein, leucocytes Tracheal secretion: Lymphocyte subpopulation, c reactive protein, lactate dehydrogenase, granulocyte macrophage colony stimulating factor, interferon γ, interleukins 10, 12 (p70), 13, 1β, 2, 4, 5, 6, 7, 8, tumor necrosis factor α
Changes in the subjective overall impairment, coughing frequency, breathlessness, mucous congestion, color of sputum, consistency of sputum on the visual analogue scale | at day 1, 3, 10 after tracheostomy
  Subjective estimation of the respiratory impairment will be analyzed via visual analogue scale (Subjective overall impairment, coughing frequency, breathlessness, mucous congestion, color of sputum, consistency of sputum).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Knopf, PD Dr., Principal Investigator — HNO, Klinikum rechts der Isar, TU München
Locations (1):
- HNO, Klinikum rechts der Isar, Technische Universität München, Munich, Bavaria, Germany

REFERENCES:
- [Background] Braun A, Steinecker M, Schumacher S, Griese M. Surfactant function in children with chronic airway inflammation. J Appl Physiol (1985). 2004 Dec;97(6):2160-5. doi: 10.1152/japplphysiol.00523.2004. Epub 2004 Aug 13. PMID 15310745
- [Background] Hofauer B, Bas M, Strassen U, Matsuba Y, Mansour N, Knopf A. [Liposomal local therapy of sinunasal symptoms in ANCA associated vasculitis]. Laryngorhinootologie. 2014 Jul;93(7):461-6. doi: 10.1055/s-0034-1372588. Epub 2014 Apr 28. German. PMID 24777579
- [Background] Hofauer B, Bas M, Manour N, Knopf A. [Liposomal local therapy as treatment for sicca symptoms in patients with primary Sjogren's syndrome]. HNO. 2013 Nov;61(11):921-7. doi: 10.1007/s00106-013-2736-x. German. PMID 23868654